CLINICAL TRIAL: NCT03672942
Title: A Proximal Change Experiment: Testing the Effects of Communication Skills Training vs. Mindfulness Techniques on Intimate Partner Aggression
Brief Title: Communication Skills vs. Mindfulness for IPV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Julia C. Babcock, Associate Professor, University of Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00000975
Record Dates: First submitted 2018-08-07; First posted 2018-09-17 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Domestic Violence; Domestic Abuse; Family Conflict; Aggression
Keywords: intimate partner violence; aggression; batterers intervention; mindfulness; communication skills; couples
MeSH Terms: conditions — Aggression | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: random assignment to two active conditions vs. a placebo control
Who Masked: Participant
Masking Description: couples are not informed as to what condition they are assigned
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Communication Skills (Experimental): Male and female participants will listen to a description of John Gottman's Gentle Start-up communication skills training exercise and practice the technique in the lab for approximately 8 minutes.
  Interventions: Behavioral: Communication Skills Training
- Mindfulness (Experimental): Male and female participants will listen to a script about Acceptance/Willingness of unwanted emotions written by Amie Zarling and practice this technique in the lab for approximately 8 minutes.
  Interventions: Behavioral: Mindfulness
- Placebo (Placebo Comparator): Male and female participants will listen to music in lieu for 8 minutes.
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Communication Skills Training — Gentle start-up is one treatment technique in the Creating Healthy Relationship Program written by John Gottman, Ph.D.
  Other Names: Gentle Start-up
  Arms: Communication Skills
Behavioral: Mindfulness — Acceptance/willingness of unwanted emotions is treatment technique of Achieving Change through Value-Based Behavior (ACTV) written by Amie Zarling, Ph.D.
  Other Names: Acceptance/Willingness of unwanted emotions
  Arms: Mindfulness
Behavioral: Placebo — Couples randomly assigned to this condition listen to music on headphones. This may be considered an active placebo as it is similar to a Time Out technique taught in battering interventions.
  Other Names: Time Out Condition
  Arms: Placebo

SUMMARY:
This tests the immediate impact of two brief interventions on couples reporting intimate partner violence using the proximal change experimental design. Couples will be randomly assigned to a mindfulness conditions, a communication exercise or a placebo condition. Outcome measures include observed and experimentally assessed aggression.

DETAILED DESCRIPTION:
This pilot study is designed to test the effects of two brief interventions on communication and emotional expression between intimate partners who have experienced recent domestic violence. In addition, it will provide some basic laboratory findings on differences in distress tolerance between perpetrators and victims of domestic abuse. Specifically, using the proximal change experimental design, couples will engaged in a 7.5 minute conflict discussion while being videotaped and having their autonomic responding monitored. Then they will be randomly assigned to one of three conditions: a communication skills training exercise, a mindfulness condition, or a placebo control. Next, ,couples will engaged in second 7.5 minute conflict discussion. It is hypothesized that those in both the communication skills training and mindfulness condition will display more positive and less aggressive behavior in their second conflict discussion as compared to their first. It is also expected that they will administer less aggression (as measured by delivery of a loud noise) to their partner after both of the active interventions. In addition, multiple measures of distress tolerance will be administered to both partners. It is expected that couples with a characterologically violent perpetrator, he or she will evidence decreased distress tolerance and the victimized partner will evidence increased distress tolerance

ELIGIBILITY:
Inclusion Criteria:

Adult co-habituating couples Reporting some violence in the past year (score > 0 on CTS2 physical abuse subscale)

Exclusion Criteria:

Homosexual couples Children under 18 non-English speakers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-09-15 (Estimated); Primary Completion 2021-09-15 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Observed aggression | 10 minutes: Change in observed behavior/emotion from first to second conflict discussion
  Specific Affect Coding System (SPAFF; Gottman, McCoy, Coan, Collier, 1996). SPAFF categorizes 16 emotions based on facial affect, vocal tone, body language, and content of speech.
TAPS aggression paradigm | 10 minutes: Change in aggression from first to second conflict discussion
  Overt aggression will be assessed using a modified version of the Taylor Aggression Paradigm (TAP; Epstein & Taylor, 1967). The TAP is an established method to study aggression in the laboratory. It is a deceptive, competitive reaction time task in which the participant competes against an "opponent" which is actually the computer program.

CONTACTS AND LOCATIONS:
Overall Officials: Julia C Babcock, Ph.D., Principal Investigator — University of Houston

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared in a data bank.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests will be reviewed by a Data Panel Review Board

REFERENCES:
- [Background] Babcock JC, Graham K, Canady B, Ross JM. A proximal change experiment testing two communication exercises with intimate partner violent men. Behav Ther. 2011 Jun;42(2):336-47. doi: 10.1016/j.beth.2010.08.010. Epub 2011 Feb 24. PMID 21496517